CLINICAL TRIAL: NCT01415193
Title: Selective Tibial Nerve Block vs Popliteal Sciatic Nerve Block in Patients Having Total Knee Arthroplasty
Brief Title: Tibial Nerve Versus Sciatic Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 09-02-002
Record Dates: First submitted 2011-08-01; First posted 2011-08-11 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2011-08

CONDITIONS: Post Operative Analgesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selective Tibial Nerve Block (Experimental)
  Interventions: Procedure: Selective Tibial Nerve block
- Control: Sciatic Nerve Block (Active Comparator)
  Interventions: Procedure: Sciatic Nerve Block

INTERVENTIONS:
Procedure: Selective Tibial Nerve block — Use of selective pain block.
  Arms: Selective Tibial Nerve Block
Procedure: Sciatic Nerve Block — Use of Sciatic Nerve Block
  Arms: Control: Sciatic Nerve Block

SUMMARY:
The purpose of this study is to analyse the ability to selectively block the posterior tibial nerve sparing the function of the common peritoneal nerve. To assess the efficacy of blocking the posterior tibial nerve will give the same post-operative pain relief after total knee surgery compared to a sciatic nerve block.

ELIGIBILITY:
Inclusion Criteria:

* total knee replacement

Exclusion Criteria:

* History of neuralgia, diabetes, pregnancy, allergy to local anesthetic solutions

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-03; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To assess if selectively blocking only the tibial nerve component of the sciatic nerve will prevent foot drop. | Upon emergence from general anesthesia and up to 48 hours in the recovery room.
  Measure frequency of foot drop in two groups and compare results.

SECONDARY OUTCOMES:
To assess if levels of pain and analgesic requirements are similar between the two groups. | 24 hours after total knee replacement surgery.
  Administer pain scale and monitor use of analgesics to compare levels two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Sinha, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States